CLINICAL TRIAL: NCT01934595
Title: Optimal Protein Supplementation for Critically Ill Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3440; SCCM Vision (Other Grant/Funding Number: SCCM Vision Grant)
Record Dates: First submitted 2013-08-29; First posted 2013-09-04 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Critical Illness
Keywords: Critically ill; Protein; Supplement; ICU; Protein synthesis
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Varying amounts of Beneprotein (Experimental): 1.5grams/kg/day, 2.0 grams/kg/day, and 2.5 grams/kg, day
  Interventions: Dietary Supplement: Beneprotein
- 1 Gram - Standard Therapy given in ICU (Active Comparator): 1 gram/kg/day of protein
  Interventions: Dietary Supplement: Beneprotein

INTERVENTIONS:
Dietary Supplement: Beneprotein — The study will compare different protein supplementation amounts to determine if increased protein supplementation in critically ill patients improves outcomes.

SUMMARY:
It is well accepted that during critical illness there is an increase in protein breakdown and loss of lean body mass. Previous studies have shown that during critical illness muscle breakdown increases dramatically. The aim of our study is to test the hypothesis that critically ill patients have improved outcomes with higher protein supplementation.

ELIGIBILITY:
Inclusion Criteria:

* • Medical or surgical patients who are admitted or transferred to the ICU with an APACHE II score greater than or equal to 18 and who are candidates for enteral nutrition within 48 hours of admission.

Exclusion Criteria:

* • Patients who cannot tolerate enteral nutrition

  * Patients who have a contraindication for enteral nutrition per American Society of Enteral and Parenteral Nutrition guidelines (GI obstruction, intractable nausea and/or vomiting, short bowel syndrome, distal GI fistula, GI bleeding that will require endoscopy, malabsorption that requires TPN, inability to access the GI tract
  * Patients with chronic stage III or IV kidney disease and/or patients receiving dialysis within six months of this hospital admission as these patients are known to require specific protein diets as an outpatient. Patients with acute kidney injury will not be excluded as there is no evidence to suggest these patients require a specific protein diet secondary to their acute kidney injury.
  * Patients with refractory hypotension unresponsive to vasoactive medications
  * Patients who are unlikely to survive the next 48 hours at the time of enrollment (this will be judged by the treating physician)
  * Patients who are unable to give consent and do not have a family member able to give consent on his/her behalf.
  * Patients with end stage liver disease or undergoing liver transplant or liver resection surgery
  * Patients whose physician thinks he/she should not participate
  * Prisoners
  * Pregnant women (all female of childbearing age will have a urine pregnancy test prior to randomization)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2017-07 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Cumulative Organ failure free days | 28 days
  The primary outcome will be cumulative organ failure free days (defined as no aggressive medical support for the patient's vital organ systems; including cardiovascular, respiratory, renal, bone marrow, and liver.

SECONDARY OUTCOMES:
Mortality | 28 days

OTHER OUTCOMES:
Number of days in ICU | 28 days
Infection Rate | 28 days
Discharge location | 28 days
New or Significantly worsening skin breakdown | 28 days
Mechanical Vent free days | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Karen S Allen, MD, Principal Investigator — OUHSC
Locations (1):
- OUHSC, Oklahoma City, Oklahoma, United States